CLINICAL TRIAL: NCT03563417
Title: International Randomized Trial on the Effect of Revascularization or Optimal Medical Therapy of Chronic Total Coronary Occlusions With Myocardial Ischemia - ISCHEMIA-CTO Trial
Brief Title: ISCHEMIA-CTO Trial - Revascularisation or Optimal Medical Therapy of CTO
Acronym: ISCHEMIA-CTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, Consultant MD PhD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISCHEMIA-CTO Trial
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Heart Disease; Chronic Total Occlusion of Coronary Artery
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI (Active Comparator)
  Interventions: Procedure: Percuteneous Coronary Intervention
- OMT (Other)
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Procedure: Percuteneous Coronary Intervention — PCI of Chronic Total Occlusions
  Arms: PCI
Other: Optimal Medical Therapy — Initiation and titration of optimal medical therapy in the control arm.
  Arms: OMT

SUMMARY:
Study design

Prospective randomized open labeled multicenter study

Hypotheses

1. In asymptomatic patients with ≥ 10% of myocardial ischemia: PCI (Percutaneous Coronary Intervention) with latest generation of drug eluting stents is superior to optimal medical therapy in terms of relative reduction in MACCE (Major Adverse Cardiovascular and Cerebrovascular events).
2. In symptomatic patients with ≥ 5% of myocardial ischemia: PCI with latest generation of drug eluting stents is superior to optimal medical therapy (OMT) in terms of improved life quality measured as an increase of SAQ (Self Assessment Questionnaire) score of 8 points after 6 months.

Inclusion Criteria

* CTO in native coronary artery
* Myocardial ischemia in a territory supplied by CTO assessed by nuclear imaging.
* Age ≥18 yrs.
* Able to provide written Informed consent and willing to comply with the specified follow-up contacts
* Target artery ≥ 2.5 mm

Prior to randomization all patients undergo 3 months of OMT. Subsequently the population will be divided into:

Cohort A: Asymptomatic (CCS < 2 and SAQ QoL > 60) patients with myocardial ischemia (≥ 10% of LV) in a territory supplied by CTO

Cohort B: Symptomatic patients (CCS class ≥ 2 and/or SAQ QoL score ≤ 60 after treating non CTO lesions and after OMT) with Myocardial ischemia (5% of LV) in a territory supplied a CTO

Cohort C: patients enrolled but not randomized in cohort A or B

Exclusion criteria (for both cohort A and B)

* NSTEMI or STEMI within 1 month
* Coronary anatomy not suitable for CTO-procedure
* Coronary artery disease involving the left main/three-vessel disease with indication for CABG following heart team conference
* Life expectancy < 2 years
* Severe chronic pulmonary disease (FEV1 < 30 % of predicted value)
* Contraindication to dual anti-platelet therapy
* Pregnancy
* eGFR < 30 mL/min/1.73 m2
* In multi-vessel disease: if it is deemed unsafe to treat the non-CTO lesion first.
* Severe valvular heart disease

Primary endpoint

Cohort A: Composite endpoint of MACCE (all-cause mortality, stroke, any myocardial infarction, clinically driven revascularization*), hospitalization for heart failure or incidence of malignant arrhythmias.

*CCS class ≥ 2 and/or QoL score < 60. Same criteria used as for allocation to Cohort B

Cohort B: SAQ Quality of Life Assessment after 6 months.

Number of patients

1,560 (1200 in cohort A/360 in cohort B

Follow up time

Cohort A: 5 years Cohort B: 6 months

DETAILED DESCRIPTION:
A chronic total occlusion (CTO) is observed in up to (1) 30 % of patients undergoing diagnostic coronary angiography. The presence of a CTO is associated with worse outcome compared to non-occlusive coronary artery disease.

Percutaneous Coronary Intervention (PCI) treatment of CTO lesions has gained much attention over the last decade due to introduction of new techniques and devices resulting in high success rates in dedicated centers. However the scientific evidence is mainly based on observational studies and expert consensus. The current European and American guidelines on revascularization does not provide any clear recommendations how to manage patients with CTO.

The indication of treating a CTO lesion, or any other lesion with PCI for that matter, is either to relieve symptoms or improve prognosis. However, to date, there are no randomized clinical trials showing any prognostic benefit from CTO revascularization. Data from randomized clinical trials are also scarce regarding improvement of symptoms and Quality of life (QoL). In the recently presented DECISION-CTO study, patients were randomized to PCI vs. OMT, and the study failed to demonstrate a prognostic or symptomatic benefit of PCI vs. OMT. However, the study was prematurely terminated due to slow inclusion rate and had a high crossover rate and a high proportion did not have a quality of life score at follow-up. The fact that both the Decision CTO and the Euro CTO trial failed to include the pre-specified number of patients, makes it difficult to draw any conclusions on how to treat these patients. The preliminary results from both trials indicate that CTO PCI seems to be a safe procedure and might improve symptoms and QoL. In the randomized EXPLORE trial, patients with ST-elevation myocardial infarction (STEMI)and a concomitant CTO in a non infarct related artery was investigated. This study showed no benefit in terms of improving left ventricular function due to CTO-PCI of the concomitant CTO, although the procedure was safe.

Meta-analysis of observational studies comparing the prognosis after successful vs. unsuccessful CTO PCI indicate prognostic and symptomatic benefit of successful CTO PCI. However, these studies often lack data regarding ischemia burden and viability. The fact that the non-successful PCI patients consistently in these studies have higher risk profile, indicating the presence of residual confounders not accounted for in the multivariate statistical models, makes the interpretation of these data in a clinical setting difficult. The non-randomized FACTOR trial demonstrated a positive outcome for quality of life, but only in symptomatic patients. Data from the OPEN-CTO registry demonstrated an improvement of the Seattle Angina Questionnaire for quality of life by 10.8 points after a successful CTO-procedure. In addition to symptomatic improvement, a successful CTO procedure can reduce the amount of myocardium susceptible to ischemia in patients with at least mild to moderate ischemia at baseline and by that the prognosis can be improved (mortality, myocardial infarction, ventricular arrhythmias).

Hence, the interventional management of CTO lesions must address whether it is indicated on symptomatic and/or prognostic basis. These questions have not been sufficiently addressed in the previous trials and we need evidence from randomized clinical trials on how to treat these patients. We therefore designed this randomized clinical trial addressing the impact of CTO PCI on outcome. Patients are included in 2 different patient cohorts depending on level of symptoms and level of myocardial ischemia. From previous studies, we know that it is most probably only patients with at least moderate myocardial ischemia who will benefit from CTO PCI in terms of improving MACCE, and only symptomatic patients who will benefit with regard to improvement of quality of life following CTO PCI.

Before entering the study all patients will be subject to a 3-month period with titration of optimal medical therapy. Hereafter the patients will be eligible for inclusion in one of two cohorts based on level of ischemia and presence of symptoms:

Cohort A: Comprise CTO patients who are asymptomatic (CCS class <2 and SAQ QoL> 60) but have moderate myocardial ischemia (>10% of the left ventricle) on MR or rubidium-PET. These patients will be randomized to CTO PCI or OMT and followed up to 10 years.

Cohort B: Comprise symptomatic CTO patients (CCS class ≥ 2 and/or SAQ QoL score ≤ 60) with at least 5% reversible ischemia. These patients will be randomized to CTO PCI or OMT. The patients randomized to OMT will be offered CTO PCI procedure 6 months after randomization following assessment of Seattle Angina Questionnaire quality of life score.

Cohort C - Patients enrolled but not eligible for randomization All patients enrolled at baseline but who do not meet the criteria described in cohort A and B for randomization. Registry based follow-up (optional) is performed at the same time points as in Cohort A.

This is the first randomized study that addresses improvement of prognosis and quality of life following PCI of CTO lesions specifically.

The purpose of this study is twofold:

1. Investigate the outcome of PCI vs. optimal medical therapy of CTO lesions in patients with significant myocardial ischemia (≥ 10%) without symptoms
2. Investigate the outcome of PCI vs. optimal medical therapy of CTO lesions in patients with symptoms and mild to moderate myocardial ischemia (≥5%).

Hypotheses

1. In asymptomatic patients with ≥ 10% of myocardial ischemia: PCI with latest generation of drug eluting stents is superior to optimal medical therapy in terms of outcome measured as 30% relative reduction in Major Adverse Cardiovascular and Cerebrovascular events (MACCE).
2. In symptomatic patients with ≥ 5% of myocardial ischemia: PCI with latest generation of drug eluting stents is superior to optimal medical therapy in terms of improved life quality measured as an increase of SAQ score of 8 points after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* CTO in native coronary artery
* Myocardial ischemia in a territory supplied by CTO assessed by nuclear imaging.
* Age ≥18 yrs.
* Able to provide written informed consent and willing to comply with the specified follow-up contacts.
* Target artery ≥ 2.5 mm

Prior to randomization all patients undergo 3 months of OMT. Subsequently the population will be divided into:

Cohort A: Asymptomatic (CCS < 2 and SAQ QoL > 60) patients with myocardial ischemia (≥ 10% of LV) in a territory supplied by CTO

Cohort B: Symptomatic patients (CCS class ≥ 2 and/or SAQ QoL score ≤ 60 after treating non CTO lesions and after OMT) with Myocardial ischemia (5% of LV) in a territory supplied a CTO assess by nuclear imaging.

Cohort C: Screening population not eligible for randomization in cohort A or B

Exclusion Criteria:

* NSTEMI or STEMI within 1 month
* Coronary anatomy not suitable for CTO-procedure
* Coronary disease involving the left main/three vessel disease with indication for CABG following heart team conference.
* Life expectancy < 2 years
* Severe chronic pulmonary disease (FEV1 < 30 % of predicted value)
* Contraindication to dual anti-platelet therapy
* Pregnancy
* eGFR < 30 mL/min/1.73 m2
* In multi-vessel disease: if it is deemed unsafe to treat the non-CTO lesion first.
* Severe valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cerebral and Cardiovascular Events | 5 Year
  Primary outcome in the Cohort A.
Quality of life - Seattle Angina Questionnaire | 6 months
  Primary outome in the Cohort B

CONTACTS AND LOCATIONS:
Overall Officials: Evald Christiansen, MD PhD, Principal Investigator — Aarhus University Hospital
Locations (27):
- Denmark (5):
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- North-Estonia Medical Centre, Tallinn, Estonia
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Heart Hospital Tampere, Tampere
  - Turku University Hospital, Turku
- France (2):
  - Clinique Louis Pasteur, Essey-lès-Nancy
  - Cardiovascular Institute, Groupe Hospitalier Mutualiste, Grenoble
- Spain (8):
  - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Galdakao, Galdakao, Bizkaia
  - Hospital Vall de Hebron, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital la Paz, Madrid
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skaane University Hospital (Lund), Lund
  - Stockholm South Central Hospital (Södersjukhuset), Stockholm
- United Kingdom (4):
  - Belfast Health and Social Care Trust, Department of Cardiology, Belfast
  - University Hospital Bristol, Bristol
  - Barts Health NHS, London
  - St George's University Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rinfret S, Sandesara PB. Reducing Ischemia With CTO PCI: Good News, But Questions Remain. JACC Cardiovasc Interv. 2021 Jul 12;14(13):1419-1422. doi: 10.1016/j.jcin.2021.05.028. No abstract available. PMID 34238552